CLINICAL TRIAL: NCT03939260
Title: The Effects of Low Flow Extracorporeal CO2 Removal on Mechanical Power in ARDS Patients
Brief Title: ECCO2R - Mechanical Power Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, Professor, University of Milan
Other Study IDs: 13175/2019
Record Dates: First submitted 2019-04-16; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: ARDS, Human; Extracorporeal CO2 Removal; Mechanical Power
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Extracorporeal CO2 Removal — Extracorporeal carbon dioxide removal (ECCO2R), a low flow extracorporeal CO2 removal, may be used in association with ultraprotective mechanical ventilation (tidal volume < 6 ml/kg and Pplat <20-25 cmH2O).

SUMMARY:
Although mechanical ventilation remains the cornerstone of ARDS treatment, several experimental and clinical studies have undoubtedly demonstrated that it can contribute to high mortality through the developing of ventilator induced lung injury even in patients with plateau pressure <30 cmH2O. Since now there are no studies exploring the application of low flow extracorporeal CO2 removal and ultraprotective ventilation to reduce mechanical power, a composite index of VILI, independently from the value of plateau pressure or the severity of hypercapnia.

ELIGIBILITY:
Inclusion Criteria:

ARDS patients undergoing mechanical ventilation with:

* PaO2/FiO2 <150 with a level of positive end expiratory pressure (PEEP) of 10 cmH2O or higher with a FiO2 > 0.5
* Plateau pressure of 28 cmH2O or higher with tidal volume of 6 ml/Kg of ideal body weight
* Mechanical power of 18 J/min or higher.

Exclusion Criteria:

* <18 years of age
* Pregnancy
* Obesity with BMI> 30
* Platelets <30 G/l
* Decompensated heart failure or acute coronary syndrome
* Acute brain injury
* Contraindication for systemic anticoagulation (for example, gastrointestinal bleeding, recent cerebrovascular accident, or chronic bleeding disorder, recent major surgery)
* Patient moribund, decision to limit therapeutic interventions
* Catheter access to femoral vein or jugular vein impossible
* Pneumothorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult respiratory distress syndrome (ARDS) patients, affected by a life-threatening condition characterized by nonhydrostatic pulmonary edema that can be caused by pulmonary (eg, pneumonia, aspiration) or nonpulmonary (eg, sepsis, pancreatitis, trauma) insults and accounts for 10% of intensive care unit (ICU) admissions. Mortality remains high ranging from 35% to 46% and it has been estimated that at least 150,000 individuals die each year of adult respiratory distress syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Mechanical Power reduction. | Changes from baseline to day 5.
  Achievement of Mechanical Power reduction under 18 J/min while maintaining pH and PaCO2 to ± 20% of baseline values obtained at tidal volume of 6 mL/kg.
  Mechanical Power (MP) (J/min) = 0.098 * respiratory rate * tidal volume (inspiratory peak airway pressure - 1/2 * (airway pressure at end inspiratory pause - airway pressure at PEEP))

SECONDARY OUTCOMES:
Respiratory mechanics. | Every six hours, every day until the fifth day or until the weaning from ECCO2R if lower than five days
  1. Respiratory system elastance (Ers) (cmH2O/L) = (airway pressure at end inspiratory pause - airway pressure at PEEP) / tidal volume
Respiratory mechanics. | Every six hours, every day until the fifth day or until the weaning from ECCO2R if lower than five days
  2. Lung elastance (El) (cmH2O/L) = (transpulmonary pressure at end inspiratory pause - transpulmonary pressure at PEEP / tidal volume
Respiratory mechanics. | Every six hours, every day until the fifth day or until the weaning from ECCO2R if lower than five days
  3. Chest wall elastance (Ecw) (cmH2O/L) = (esophageal pressure at end inspiratory pause - esophageal pressure at PEEP) / tidal volume
Respiratory mechanics. | Every six hours, every day until the fifth day or until the weaning from ECCO2R if lower than five days
  4. End inspiratory transpulmonary pressure (cmH2O)= airway pressure at end inspiratory pause - (esophageal pressure at end inspiratory pause - expiration at atmospheric pressure by a release manouvre).
Gas exchange. | Every six hours, every day until the fifth day or until the weaning from ECCO2R if lower than five days
  Assessment of changes in PaCO2 mmHg.
Gas exchange. | Every six hours, every day until the fifth day or until the weaning from ECCO2R if lower than five days
  Assessment of changes in PaO2 mmHg.
Gas exchange. | Every six hours, every day until the fifth day or until the weaning from ECCO2R if lower than five days
  Assessment of changes in PaO2/FiO2.
Safety assessment and adverse device related events: frequency of serious adverse events | Every day, until the fifth day or until the weaning from ECCO2R if lower than five days
  Safety assessment reporting frequency of serious adverse events in terms of device related mechanical events (Pump malfunction, membrane lung clotting, system leaks, tubing rupture, air in the circuit) and device related clinical events (heamolysis, significant bleeding, thromboembolic complications, neurologic complications, metabolic complications).

CONTACTS AND LOCATIONS:
Locations (1):
- ASST-Santi Paolo e Carlo, San Paolo Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Fan E, Needham DM, Stewart TE. Ventilatory management of acute lung injury and acute respiratory distress syndrome. JAMA. 2005 Dec 14;294(22):2889-96. doi: 10.1001/jama.294.22.2889. PMID 16352797
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Chiumello D, Brochard L, Marini JJ, Slutsky AS, Mancebo J, Ranieri VM, Thompson BT, Papazian L, Schultz MJ, Amato M, Gattinoni L, Mercat A, Pesenti A, Talmor D, Vincent JL. Respiratory support in patients with acute respiratory distress syndrome: an expert opinion. Crit Care. 2017 Sep 12;21(1):240. doi: 10.1186/s13054-017-1820-0. PMID 28899408
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367
- [Background] Kolobow T, Gattinoni L, Tomlinson T, Pierce JE. An alternative to breathing. J Thorac Cardiovasc Surg. 1978 Feb;75(2):261-6. PMID 625133
- [Background] Peek GJ, Clemens F, Elbourne D, Firmin R, Hardy P, Hibbert C, Killer H, Mugford M, Thalanany M, Tiruvoipati R, Truesdale A, Wilson A. CESAR: conventional ventilatory support vs extracorporeal membrane oxygenation for severe adult respiratory failure. BMC Health Serv Res. 2006 Dec 23;6:163. doi: 10.1186/1472-6963-6-163. PMID 17187683